CLINICAL TRIAL: NCT03754426
Title: Validation of MolecuLight Phoenix Prototypes in Clinic
Brief Title: A Prospective, Pilot Evaluation of Device Equivalence
Acronym: Equivalence
Status: Completed | Type: Observational
Sponsor: MolecuLight Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 18-009
Record Dates: First submitted 2018-11-22; First posted 2018-11-27 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Wound
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Fluorescence Imaging Device — Hand-held, real-time fluorescence imaging device

SUMMARY:
Patients with chronic wounds will be imaged using 3 imaging devices. Two types of images will be acquired with each device, as standard photograph (ST-image) and a fluorescence image (FL-image). The images captured with the 3 imaging devices will be compared off-line by 5 interpreters to assess for any differences in the images that would alter a clinical decision.

DETAILED DESCRIPTION:
Patients (n = 50) with chronic wounds will be imaged using 3 imaging devices. Two types of images will be acquired with each device, as standard photograph (ST-image) and a fluorescence image (FL-image). The images captured with the 3 imaging devices will be compared off-line by 5 interpreters to assess for any differences in the images that would alter a clinical decision.

ELIGIBILITY:
Inclusion Criteria:

* Subjects (inpatient/outpatient) presenting with a wound
* Wound size less than 15 cm in length
* 18 years or older

Exclusion Criteria:

* Treatment with an investigational drug within 1 month before study enrolment
* Subjects with recent (<30 days) biopsy or curettage of target wound
* Subjects with wounds that cannot be completely imaged by study device due to anatomic location
* Unable or unwilling to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with chronic wounds
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2019-01-02 (Actual); Study Completion 2019-01-02 (Actual)

PRIMARY OUTCOMES:
Concordance | 2 months
  Estimate concordance of moderate/heavy bacterial load present in images acquired with each of 3 devices

CONTACTS AND LOCATIONS:
Overall Officials: Ron Linden, MD, Principal Investigator — Judy Dan Research and Treatment Centre
Locations (1):
- Judy Dan Research and Treatment Centre, North York, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to disseminate information to patients. If patients ask for their information then they will be provided a response with the most up to date information.